CLINICAL TRIAL: NCT03796871
Title: Interest of a New Medical Device for the Visualization of Cutaneous Lesions Based on Polarized Light
Brief Title: Medical Device Based on Polarized Light for Cutaneous Lesions Visualization
Acronym: DERMAPOL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: not enough patients
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 6798
Record Dates: First submitted 2018-12-06; First posted 2019-01-08 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Skin Lesion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dermapol (Experimental): Use of the experimental medical device
  Interventions: Device: Dermapol

INTERVENTIONS:
Device: Dermapol — Use of the experimental medical device before lesion excision : skin lesion lighting (4 wavelengths) for less than 1 minute and image recording

SUMMARY:
Skin cancers represent a real public health issue. The diagnosis of pre-cancerous lesions thus is a priority. The diagnosis gold standard is based on the combination of clinical and histopathological examinations. Nevertheless, the clinical examination is not sufficiently effective, meaning that a biopsy has to be done for each suspected lesion. In order to avoid unnecessary biopsy excisions, a new medical device (DERMAPOL) was designed to help dermatologists in diagnosing skin lesions.

This medical device combined with its software is a strong and ergonomic spectro-polarimetric imager instrument. It can realize images of the superficial cutaneous tissues and subcutaneous tissues close to the surface by exploiting polarized light properties.

This first clinical trial aims to demonstrate that this medical device is able to segment effectively healthy and tumor tissues and that it can correlate main semiological elements (identified thanks to the clinical and histopathological examinations) to the physico-optical characteristics obtained on the images of the medical device.

ELIGIBILITY:
Inclusion Criteria:

* adult patient with a skin tumor (benign or cancerous) which has to be excised and analysed according to histopathological examination
* skin lesion belonging to one of these groups (diagnosed by clinical examination):

  * cutaneous cyst
  * seborrhoeic keratosis
  * cutaneous carcinoma
  * naevus
  * melanoma
  * actinic keratosis and cutaneous horn
  * other skin tumors
* skin lesion size equal to or less than 5 cm
* signed written consent form
* patient affiliated to a social insurance

Exclusion Criteria:

* skin lesion size strictly over than 5 cm
* eyelid lesion
* aluminium, POM (polyoxymethylene) or organic glass allergy
* known pregnancy, breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2024-01-14 (Actual); Study Completion 2024-01-14 (Actual)

PRIMARY OUTCOMES:
Proportion of lesions with semiological characteristics | Before biopsy
  Proportion of lesions for which at least one semiological characteristic (detected by the combination of visual and histopathological examinations) was identified by the medical device thanks to physico-optical properties

SECONDARY OUTCOMES:
Physico-optical description of the lesions | Before biopsy
  Physico-optical description of the cutaneous lesions by the medical device
Number of different semiological characteristics | Before biopsy
  Number of different semiological characteristics visualized by the medical device and by the combination of clinical and histopathological examinations for each image processing
Proportion of semiological characteristics properly identified | Before biopsy
  Proportion of semiological characteristics properly identified by the medical device for all lesions
Specificity, sensitivity and predictive values | Before biopsy
  Specificity, sensitivity, true positive rate, true negative rate, false positive rate, false negative rate of the medical device, for each semiological characteristic identified by the combination of the clinical and histopathological examinations
Cases proportion for which the same semiological characteristics list was found between the medical device and the combination of clinical and histopathological diagnosis | Before biopsy
  Proportion of cases with same semiological characteristics list

CONTACTS AND LOCATIONS:
Overall Officials: Bernard CRIBIER, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No